CLINICAL TRIAL: NCT04478864
Title: Assessment of Knowledge, Practice and State of Periodontal Health Among Egyptian Patients Attending Diagnostic Center at Faculty of Dentistry, Cairo University. A Cross-sectional Study
Brief Title: Knowledge, Practice and State of Periodontal Health
Status: Completed | Type: Observational
Sponsor: Noha Ayman Ghallab (Other)
Responsible Party: Sponsor-Investigator, Noha Ayman Ghallab, Prof. Dr Noha Ayman Ghallab - Professor of Oral Medicine and Periodontology / Cairo University., Cairo University
Organization: Cairo University (Other)
Other Study IDs: Esraa2020
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to assess the knowledge and practice of periodontal health, which will be done using a well constructed and validated questionnaire. Then periodontal health status of all participants will be assessed via clinical examination of certain teeth.

DETAILED DESCRIPTION:
The primary outcome of the study is the knowledge of periodontal health.It will be assessed by 10 questions focusing on the basic knowledge of gingival appearance, causes and consequence of periodontal disease, impact of systemic disease on the progression of periodontal conditions, and prevention. Then, periodontal practice will be addressed via several questions that evaluate the self-care practices of tooth brushing, flossing, mouth rinsing in recent one year, scaling in recent five years, and how to alleviate gingival bleeding if there is.

Periodontal examination using the community periodontal index (CPI) will be done for all of the participants to assess the status of periodontal condition. The dentition will be divided into sextants and the highest code number corresponding to the worst periodontal condition around each of the 10 indexed teeth being recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is above 15 years old.
2. Patient consulting in the outpatient clinic
3. Provide informed consent.

Exclusion Criteria:

1. Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
2. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of periodontal health | "through study completion, an average of 1 year"
  will be assessed from the 10 questions in the questionnaire and be presented as frequencies and percentages.

SECONDARY OUTCOMES:
Periodontal health practice | "through study completion, an average of 1 year"
  Five questions regarding practice will be analyzed and presented as frequencies and percentages
State of periodontal health | "through study completion, an average of 1 year"
  will be determined by measuring the community periodontal index of treatment needs (CPITN) and modified community periodontal index (CPI) that measures the clinical attachment level (CAL) scores, both giving a score of zero to the best periodontal condition and a score of 4 to the worst one

CONTACTS AND LOCATIONS:
Overall Officials: Noha A Ghallab, MD, Study Director — Professor of Oral Medicine and Periodontology, Cairo University
Locations (1):
- Faculty of Oral & Dental Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murakami S, Mealey BL, Mariotti A, Chapple ILC. Dental plaque-induced gingival conditions. J Periodontol. 2018 Jun;89 Suppl 1:S17-S27. doi: 10.1002/JPER.17-0095. PMID 29926958
- [Background] Gronbeck Linden I, Hagglin C, Gahnberg L, Andersson P. Factors Affecting Older Persons' Ability to Manage Oral Hygiene: A Qualitative Study. JDR Clin Trans Res. 2017 Jul;2(3):223-232. doi: 10.1177/2380084417709267. Epub 2017 May 15. PMID 30938636
- [Background] Holtzman JS, Atchison KA, Macek MD, Markovic D. Oral Health Literacy and Measures of Periodontal Disease. J Periodontol. 2017 Jan;88(1):78-88. doi: 10.1902/jop.2016.160203. Epub 2016 Aug 13. PMID 27523517